CLINICAL TRIAL: NCT02471781
Title: Zenith® TX2® Low Profile TAA Endovascular Graft Clinical Study
Brief Title: Zenith® TX2® Low Profile TAA Endovascular Graft
Status: Approved for marketing | Type: Expanded Access
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-001 CA; NCT02319551 (obsolete NCT alias)
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Aortic Aneurysm; Penetrating Ulcer; Vascular Disease
Keywords: Aortic Aneurysm; Aneurysm; Vascular Prosthesis; Vascular Disease; Blood Vessel Prosthesis Implantation
MeSH Terms: conditions — Aortic Aneurysm; Penetrating Atherosclerotic Ulcer; Vascular Diseases; Aneurysm

INTERVENTIONS:
Device: Zenith TX2 Low Profile TAA Endovascular Graft — Endovascular treatment of patients with aneurysms or ulcers of the descending thoracic aorta having morphology suitable for endovascular repair.
  Other Names: Zenith Alpha Thoracic™ Endovascular Graft

SUMMARY:
The Zenith TX2 Low Profile TAA Endovascular Graft extended study is to collect confirmatory safety and effectiveness data. The Zenith TX2 Low Profile TAA Endovascular Graft is indicated for the treatment of patients with a descending thoracic aortic aneurysm or penetrating ulcer and has an anatomy suitable for repair.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following

  * Descending thoracic aneurysm with diameter ≥ 5.0 cm
  * Descending thoracic aneurysm with a history of growth ≥ 0.5 cm per year
  * Descending thoracic degenerative or atherosclerotic ulcer ≥ 10 mm in depth and 20 mm in diameter

Exclusion Criteria:

* Life expectancy less than 2 years
* Pregnant of breastfeeding or planning on becoming pregnant within 60 months
* Unwilling to comply with the follow-up schedule
* Less than 30 days beyond primary endpoint for other investigative drug or device study
* Receiving home oxygen
* Myocardial infarction within the last 3 months
* Stroke within the last 3 months
* Diagnosed or suspected congenital degenerative collagen disease
* Systemic infection
* Bleeding diathesis, uncorrectable coagulopathy, or refuses blood transfusion
* Allergy to polyester, polypropylene, nitinol, or gold
* Previous placement of a thoracic endovascular graft
* Prior open repair involving the descending thoracic aorta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Karl Illig, MD, Principal Investigator — Dialysis Access Center
Locations (15):
- United States (15):
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Indiana Heart Hospital, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Mount Sinai Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania